CLINICAL TRIAL: NCT04410315
Title: Elevated Serum-lactate in Patients With Brain Tumor During and After Elective Craniotomy: an Observational Clinical Study of Postoperative Patient Outcome.
Brief Title: Hyperlactatemia During and After Tumorcraniotomy
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Alexandra Vassilieva, Principal investigator, Rigshospitalet, Denmark
Other Study IDs: Prosp.Laktat.Tumorkraniotomi
Record Dates: First submitted 2020-05-14; First posted 2020-06-01 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Hyperlactatemia; Brain Tumor; Surgery; Anesthesia
MeSH Terms: conditions — Hyperlactatemia; Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tumorcraniotomy patients
  Interventions: Other: Serum-lactate < 2,2 mmol/L; Other: Serum-lactate >/= 2,2 mmol/L

INTERVENTIONS:
Other: Serum-lactate < 2,2 mmol/L — Bloodgas analysis every hour from start surgery until recovery ward discharge
Other: Serum-lactate >/= 2,2 mmol/L — Bloodgas analysis every hour from start surgery until recovery ward discharge

SUMMARY:
This study aims to investigate the association between hyperlactatemia and neurological disability, length-of-stay and mortality in patients who undergo tumorcraniotomy. The risk factors that induce lactat accumulation will also be explored.

DETAILED DESCRIPTION:
Hyperlactatemia is a frequent occurrence in brain tumor surgery. The existing studies, however, are all retrospective, reporting varying effects on clinical outcome. One study reported new neurological deficitis, some found an association with extended hospital stay, while others found no association with outcome. It is therefore important to conduct a prospective study of hyperlactatemia in this patientgroup.

Participants in this study will follow the standard treatment protocol for tumorcraniotomy, aside from 2-3 additional, perioperative blodgas analyses and 2 standardized measurements of neurological disability.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Must undergo elective tumor craniotomy
* Understand oral and written Danish

Exclusion Criteria:

* Adults with incapacity
* Stereotactic biopsy
* Lack of informed and signed consent to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing tumorcraniotomy
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Neurological disability | Change from baseline mRS at 30 days after surgery
  Modified Rankin Scale (Scoring 0-6, high scores meaning worse outcome)

SECONDARY OUTCOMES:
Length of hospital stay | 1 year
  In days from admission to discharge.
Mortality | After 30 days, 6 months and 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neuroanesthesiology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided